CLINICAL TRIAL: NCT04806087
Title: Validity And Reliability Of A New Method To Measure Cervical Proprioception
Brief Title: A New Method To Measure Cervical Proprioception
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Kaya Mutlu, PT, Assoc. Prof. Dr., Istanbul University - Cerrahpasa
Other Study IDs: 2019/10
Record Dates: First submitted 2021-03-14; First posted 2021-03-19 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Proprioception; Position Sense
Keywords: reliability; validity; cervical; proprioception; rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate cervical proprioception (CP), frontal plane target platforms defined Revel technique measurement commonly used as an alternative to the Cervical Range of Motion (CROM) device in laser measurements for the head repositioning accuracy (HRA) test. However, when evaluating CP, the plane where the movement of the atlanto-axial joint takes place is the horizontal plane. Therefore, the investigators aimed to investigate the validity and reliability of CP measurements conducted via AOS PropPoint® device on the horizontal and frontal platforms, and the investigators hypothesized that horizontal platform measurement is more reliable and valid than frontal plane measurement.

DETAILED DESCRIPTION:
It has been reported in a number of studies that methods utilizing laser are practical, easy, portable, and inexpensive in clinical use, a standardized and branded laser apparatus and system have not been identified. This has caused problems about whether the laser equipment used in the literature is valid and reliable in the evaluation of cervical proprioception (CP). Besides, the head repositioning accuracy (HRA) test, which was designed before for CP assessment and standardized with trigonometric equations, carries out measurements in the frontal plane. In addition, cervical rotation in the atlanto-axial joint occurs in the horizontal plane. Therefore, the investigators presume that evaluating the biomechanical motion occurring in the horizontal plane and transferring it directly to the horizontal plane will be more practical and reliable for practitioners.

The subjects' HRA values were measured through AOS ProPoint® device in the horizontal and frontal platforms and also through the CROM device. Each measurement was repeated bilaterally three times, and they were averaged. To validate the measurement method, a comparison between the CROM device used as the gold standard and the measurement values was made. Test-retest and inter-rater reliability scores were calculated to evaluate the reliability of the horizontal measurement method.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 35 years
* bilateral cervical rotation of 30 degrees and above
* being a volunteer.

Exclusion Criteria:

* all kinds of orthopedic and neurological problems that might cause head, eye and neck movement limitation; having a pacemaker, platinum, dental braces, etc., which might affect the magnetic field; and the presence of epilepsy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample consist of volunteer, healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Horizontal Plane Target Platform Measurement with AOS PropPoint® Device | Baseline
  AOS PropPoint® is a practical, easy-to-use and low-cost device designed by physiotherapists to evaluate and improve the proprioceptive senses of various joints in the body. The fabric used to attach the laser apparatus to the head is made of a special veltec fabric. The laser pointer was placed at the center of the participants' atlanto-axial joint. The laser cursor was positioned at an angle of approximately 45° with the ground and projected onto a fixed semicircular horizontal target platform drawn with intervals of one degree. It was noted that the NHP and the 0° (zero point of the horizontal plane on the ground correspond to each other. The HRA measurement of AOS PropPoint® device on the horizontal platform was made simultaneously with the CROM. The deviation of the laser pointer from 0° (zero point) on the horizontal platform was recorded.

SECONDARY OUTCOMES:
Frontal Plane Target Platform Measurement with AOS PropPoint® Device | Baseline
  Target board was improved based on the formula tang^(-1) [error distance/90 cm]. The readings was accurate to ±0.5. We also used a target platform board with a diameter of 40 cm and graded at 1 cm intervals. The laser cursor was fixed with the help of veltec fabric in the center of the frontal bone of the volunteers. The subjects were seated 90 cm away from the frontal plane for the HRA test. When the volunteers felt that they were coming back to the starting point, the amount of deviation from the starting point was recorded by asking them to give a signal by simply extending their right index finger slightly, without opening their eyes.
Cervical Proprioception assesment with Cervical Range of Motion Device (CROM) | Baseline
  The CROM device has been proven to be a reliable and valid tool for HRA tests. The volunteers were seated in a chair without back support with their knees and hip joints positioned at 90 degrees, and their left shoulders pointing to the north of the room, where the measurement was made. They were also asked to wear magnetic collars so that their left shoulders always pointed north. A subject was blindfolded and seated on a chair with their head in the neutral head position (NHP), and was asked to relocate their head on the trunk as accurately as possible after cervical rotations of 30 degrees to the left and right sides. Three trials were carried out after a right head rotation and another three after a left head rotation and they were averaged for each side. The accuracy of head repositioning was measured through the absolute value of the constant error. Randomization was achieved by randomizing the measurements starting from the right or left side.
Horizontal Plane Target Platform Measurement with AOS PropPoint® Device | Within a 5-to-7-day period after the first assessment
  AOS PropPoint® is a practical, easy-to-use and low-cost device designed by physiotherapists to evaluate and improve the proprioceptive senses of various joints in the body. The fabric used to attach the laser apparatus to the head is made of a special veltec fabric. The laser pointer was placed at the center of the participants' atlanto-axial joint. The laser cursor was positioned at an angle of approximately 45° with the ground and projected onto a fixed semicircular horizontal target platform drawn with intervals of one degree. It was noted that the NHP and the 0° (zero point of the horizontal plane on the ground correspond to each other. The HRA measurement of AOS PropPoint® device on the horizontal platform was made simultaneously with the CROM. The deviation of the laser pointer from 0° (zero point) on the horizontal platform was recorded.
Frontal Plane Target Platform Measurement with AOS PropPoint® Device | Within a 5-to-7-day period after the first assessment
  Target board was improved based on the formula tang^(-1) [error distance/90 cm]. The readings was accurate to ±0.5. We also used a target platform board with a diameter of 40 cm and graded at 1 cm intervals. The laser cursor was fixed with the help of veltec fabric in the center of the frontal bone of the volunteers. The subjects were seated 90 cm away from the frontal plane for the HRA test. When the volunteers felt that they were coming back to the starting point, the amount of deviation from the starting point was recorded by asking them to give a signal by simply extending their right index finger slightly, without opening their eye.
Cervical Proprioception assesment with Cervical Range of Motion Device (CROM) | Within a 5-to-7-day period after the first assessment
  The CROM device has been proven to be a reliable and valid tool for HRA tests. The volunteers were seated in a chair without back support with their knees and hip joints positioned at 90 degrees, and their left shoulders pointing to the north of the room, where the measurement was made. They were also asked to wear magnetic collars so that their left shoulders always pointed north. A subject was blindfolded and seated on a chair with their head in the neutral head position (NHP), and was asked to relocate their head on the trunk as accurately as possible after cervical rotations of 30 degrees to the left and right sides. Three trials were carried out after a right head rotation and another three after a left head rotation and they were averaged for each side. The accuracy of head repositioning was measured through the absolute value of the constant error. Randomization was achieved by randomizing the measurements starting from the right or left side.

CONTACTS AND LOCATIONS:
Overall Officials: Aygül Köseoğlu, PT, Study Chair — Bahçeşehir University; Ebru K Mutlu, Principal Investigator — İstanbul University- Cerrahpasa; Dilber Çoskunsu, Study Director — Bahçeşehir University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Revel M, Andre-Deshays C, Minguet M. Cervicocephalic kinesthetic sensibility in patients with cervical pain. Arch Phys Med Rehabil. 1991 Apr;72(5):288-91. PMID 2009044
- [Background] Roren A, Mayoux-Benhamou MA, Fayad F, Poiraudeau S, Lantz D, Revel M. Comparison of visual and ultrasound based techniques to measure head repositioning in healthy and neck-pain subjects. Man Ther. 2009 Jun;14(3):270-7. doi: 10.1016/j.math.2008.03.002. Epub 2008 Jun 2. PMID 18514016
- [Background] Chen X, Treleaven J. The effect of neck torsion on joint position error in subjects with chronic neck pain. Man Ther. 2013 Dec;18(6):562-7. doi: 10.1016/j.math.2013.05.015. Epub 2013 Jun 26. PMID 23810427
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238